CLINICAL TRIAL: NCT06779825
Title: Impact of Stimulants and In-Scanner Motion on FMRI Neurofeedback and Task Performance in ADHD
Brief Title: Impact of Stimulants and In-Scanner Motion on Attentive Task Performance in ADHD (ADHD_NFB)
Acronym: ADHD_NFB
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alexander Cohen, Principal Investigator and Medical Physician, Boston Children's Hospital
Other Study IDs: IRB-P00049401
Record Dates: First submitted 2025-01-09; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: ADHD
Keywords: ADHD; Neurofeedback; fMRI; attention tasks; motion
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Stimulant Medication for ADHD: Arm 1 will require that all participants refrain from taking their usual ADHD stimulant medication on the day of at least two of the study visits, one of which includes neurofeedback. Participants may resume their medication regimen upon completion of the study visit.
  Interventions: Combination Product: fMRI Neurofeedback attention task

INTERVENTIONS:
Combination Product: fMRI Neurofeedback attention task — Neurofeedback is an attentive task where participants are shown their real-time brain signals while in the scanner with the use of a representation, such as a rocket moving towards a portal. Participants are able to increase this brain signal by more purposefully engaging certain brain regions, and this is reflected in the representation that they see. Ultimately, this study is interested in whether neurofeedback can replicate the effects of stimulant medication in ADHD.

SUMMARY:
The goal of this interventional study is to learn the effects that stimulant medication prescribed to ADHD individuals has in their performance of attentive tasks, as measured by images and data collected through neuroimaging (fMRI) while also implementing new motion-correcting software. The main questions it aims to answer are:

1. How do the use of stimulants affect brain activity and motion in fMRI research in ADHD studies?
2. Can neurofeedback, an attentive task using real-time brain activity, engage the same brain circuits as seen with stimulant medication in individuals with ADHD?

Researchers will compare participant's brain activity from the completion of attentive tasks performed in the scanner while following their regular medication regimen and while abstaining to take medication. Researchers will also compare how the data collected using a more precise motion correction software differs to other previously reported data from ADHD studies who possibly employed more lenient measures of motion correction.

Participants will:

1. Be asked to complete at least 4 fMRI sessions, two of which will include neurofeedback
2. Be asked to abstain from taking stimulant medication on the day of two of these fMRI visits
3. Complete attentive tasks while in the scanner that will activate target brain regions of interest

ELIGIBILITY:
Inclusion Criteria:

* Age 12 or older
* Able to follow verbal and written instructions in native language
* Pre-existing clinical ADHD diagnosis (with or without comorbid anxiety diagnoses)
* Pre-existing medication regimen of methylphenidate or amphetamine salt derivatives with no changes in the last month

Exclusion Criteria:

* Known visual impairment preventing test administration
* Contraindication of inability to participate in fMRI scanning (per MRI screening form)
* Known, self-reported non-incidental structural brain abnormality
* Autism Spectrum Disorder or Obsessive-Compulsive Disorder
* Non-verbal

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will be largely recruited through the Boston Children Hospital's resources, such as a participant registry or from clinical practice, only applicable to individuals who fit the eligibility criteria listed above.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Neurofeedback mimicking the effects of stimulants | Through data collection and analysis, an average of 1 year
  Compare whether neurofeedback can mimic the effects of stimulants by engaging similar attentive brain circuits and providing a normalized activation effect similar to that of stimulants (measured in units of neural activation, with intensity based on p-value of significance, and by a z-score obtained in real-time during the task). This data will be collected during the completion of the neurofeeback task while in the scanner.
Performance on Attentive Tasks | Through data collection and analysis, an average of 1 year
  Performance on other attentive tasks (e.g., reaction time in seconds, accuracy of response), different from neurofeedback, will be observed while on stimulant medication, compared to performance on the same tasks while refraining from stimulant medication.
Precise motion correction as a better accountant of ADHD mechanisms | Through data collection and analysis, an average of 1 year
  Will compare results from data collected using fMRI and a new software that more precisely corrects for motion artifacts in a slice-by-slice manner to results previously reported for ADHD studies using more lenient fMRI motion artifact measures. Some of these comparisons will include more or less brain activation of the same regions, more precise windows of activation, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital @2BP, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hein IM, De Vries MC, Troost PW, Meynen G, Van Goudoever JB, Lindauer RJ. Informed consent instead of assent is appropriate in children from the age of twelve: Policy implications of new findings on children's competence to consent to clinical research. BMC Med Ethics. 2015 Nov 9;16(1):76. doi: 10.1186/s12910-015-0067-z. PMID 26553304
- [Background] Isles AF. Understood consent versus informed consent: a new paradigm for obtaining consent for pediatric research studies. Front Pediatr. 2013 Nov 21;1:38. doi: 10.3389/fped.2013.00038. PMID 24400284
- [Background] Sulzer J, Haller S, Scharnowski F, Weiskopf N, Birbaumer N, Blefari ML, Bruehl AB, Cohen LG, DeCharms RC, Gassert R, Goebel R, Herwig U, LaConte S, Linden D, Luft A, Seifritz E, Sitaram R. Real-time fMRI neurofeedback: progress and challenges. Neuroimage. 2013 Aug 1;76:386-99. doi: 10.1016/j.neuroimage.2013.03.033. Epub 2013 Mar 27. PMID 23541800
- [Background] Wu ZM, Bralten J, An L, Cao QJ, Cao XH, Sun L, Liu L, Yang L, Mennes M, Zang YF, Franke B, Hoogman M, Wang YF. Verbal working memory-related functional connectivity alterations in boys with attention-deficit/hyperactivity disorder and the effects of methylphenidate. J Psychopharmacol. 2017 Aug;31(8):1061-1069. doi: 10.1177/0269881117715607. Epub 2017 Jun 28. PMID 28656805
- [Background] Berberat J, Huggenberger R, Montali M, Gruber P, Pircher A, Lovblad KO, Killer HE, Remonda L. Brain activation patterns in medicated versus medication-naive adults with attention-deficit hyperactivity disorder during fMRI tasks of motor inhibition and cognitive switching. BMC Med Imaging. 2021 Mar 19;21(1):53. doi: 10.1186/s12880-021-00579-3. PMID 33740903
- [Background] Rubia K, Alegria AA, Cubillo AI, Smith AB, Brammer MJ, Radua J. Effects of stimulants on brain function in attention-deficit/hyperactivity disorder: a systematic review and meta-analysis. Biol Psychiatry. 2014 Oct 15;76(8):616-28. doi: 10.1016/j.biopsych.2013.10.016. Epub 2013 Oct 24. PMID 24314347
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Fair DA, Nigg JT, Iyer S, Bathula D, Mills KL, Dosenbach NU, Schlaggar BL, Mennes M, Gutman D, Bangaru S, Buitelaar JK, Dickstein DP, Di Martino A, Kennedy DN, Kelly C, Luna B, Schweitzer JB, Velanova K, Wang YF, Mostofsky S, Castellanos FX, Milham MP. Distinct neural signatures detected for ADHD subtypes after controlling for micro-movements in resting state functional connectivity MRI data. Front Syst Neurosci. 2013 Feb 4;6:80. doi: 10.3389/fnsys.2012.00080. eCollection 2012. PMID 23382713
- [Background] Dziemian S, Baranczuk-Turska Z, Langer N. Association between attention-deficit/hyperactivity disorder symptom severity and white matter integrity moderated by in-scanner head motion. Transl Psychiatry. 2022 Oct 6;12(1):434. doi: 10.1038/s41398-022-02117-3. PMID 36202807
- [Background] Couvy-Duchesne B, Ebejer JL, Gillespie NA, Duffy DL, Hickie IB, Thompson PM, Martin NG, de Zubicaray GI, McMahon KL, Medland SE, Wright MJ. Head Motion and Inattention/Hyperactivity Share Common Genetic Influences: Implications for fMRI Studies of ADHD. PLoS One. 2016 Jan 8;11(1):e0146271. doi: 10.1371/journal.pone.0146271. eCollection 2016. PMID 26745144
- [Background] Makowski C, Lepage M, Evans AC. Head motion: the dirty little secret of neuroimaging in psychiatry. J Psychiatry Neurosci. 2019 Jan 1;44(1):62-68. doi: 10.1503/jpn.180022. PMID 30565907
- [Background] Yakupov R, Lei J, Hoffmann MB, Speck O. False fMRI activation after motion correction. Hum Brain Mapp. 2017 Sep;38(9):4497-4510. doi: 10.1002/hbm.23677. Epub 2017 Jun 5. PMID 28580597
- See also: Lab website giving a brief description of study protocol for those interested in participating. — https://bchcohenlab.com/participate/neurofeedback.html